CLINICAL TRIAL: NCT02521584
Title: Ischemia Time and Graft Survival
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: AlRefaey Kandeel (Other)
Responsible Party: Sponsor-Investigator, AlRefaey Kandeel, Dr, Mansoura University
Organization: Mansoura University (Other)
Other Study IDs: Adel/2015
Record Dates: First submitted 2015-08-09; First posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Liver Transplant
Keywords: Liver transplant recipient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Study the effect of ischemia time on patient and graft survival.

DETAILED DESCRIPTION:
Study the effect of cold ischemia and warm ischemia on graft function after one year and patient one year survival.

ELIGIBILITY:
Inclusion Criteria:

* recipients of living donor liver transplantation

Exclusion Criteria:

* early mortality

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: recipients of living donor liver transplantation
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
one year graft survival | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura university, Al Mansurah, Dakahlia Governorate, Egypt